CLINICAL TRIAL: NCT05222958
Title: Effectiveness of an App for Tobacco Cessation in Pregnant Women
Brief Title: Effectiveness of an App for Tobacco Cessation in Pregnant Women (TOBBGEST)
Acronym: TOBBGEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4R21/134
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-03

CONDITIONS: Pregnant Women
Keywords: Tobacco; Pregnant women; Gamification; Telemedicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: (Experimental): The intervention consists of using a smoking cessation app. Patients assigned to the intervention group will be given the access code to the Gestobb App and advice on how to use it.
  Interventions: Device: Gestob App
- No intervention (No Intervention): Patients in the control group will continue their follow-up visits at ASSIR and will be offered smoking cessation treatment following standard practice protocols.

INTERVENTIONS:
Device: Gestob App — Gestop App is a mobile app that aims to help pregnant women quit smoking through gamification. It also allows you to obtain information about tobacco and pregnancy.
  Arms: Experimental:

SUMMARY:
Background: Tobacco use during pregnancy is one of the most modifiable causes of morbidity and mortality for both pregnant women and their fetus. Despite the fact that smoking among pregnant has decreased in recent years, smoking continues to be a major public health problem.

Hypothesis / Research question: The use of new technologies such as applications (apps) for mobile devices designed with a gamification strategy (understood as an incentive through play) could help women to quit smoking during pregnancy and in the long term. A structured App-based intervention using gamification adapted to pregnant women will decrease smoking prevalence in this population.

Objectives: To evaluate the effectiveness of an intervention against tobacco in pregnant women based on an app for tobacco abstinence. Specific objectives: 1) To determine the effectiveness of the intervention on smoking cessation during pregnancy, 2) Determine the effectiveness of the intervention in in the long term and 3) To determine the impact of the intervention to reduce smoking in pregnant women who continue smoking.

Design: Randomized, multicentre community intervention trial

Setting: Sexual and Reproductive Health Care Services of the Camp de Tarragona and Central Catalonia Primary Care Centres.

Intervention: the participants will have the usual clinical practice intervention and the intervention group (IG) will also have access to an app based on gamification, verified by coximetry during the follow-up, and with a cotinine test at the end.

Analysis: of groups "by intention to treat", abstinence rates will be compared and the determining factors will be evaluated using multivariate statistics.

Expected results: smoking cessation in the IG will be > 5%, compared to normal practice.

Applicability and Relevance: It promotes activities aimed to reduce tobacco consumption in the general population, and especially in women, in order to decrease comorbidity associated with long-term smoking, which will lead to a reduction in tobacco-related diseases in the whole population.

DETAILED DESCRIPTION:
Design: community-based intervention trial with simple random assignment.

Setting and study population: the study population will be drawn from the usual consultations of 4 Sexual and Reproductive Health Care Centres (ASSIR) responsible for pregnancy monitoring in the community, managed by the Catalan Health Institute (ICS) in Tarragona and Barcelona.

Study subjects: pregnant women over 18 years of age who attended the ASSIR services and consented to participate in the study and meet the inclusion criteria.

Randomisation process of the intervention: the participants included will be assigned to receive or not to receive the proposed intervention. The allocation sequence will be carried out consecutively, centralised from the Research Support Unit of the Jordi Gol Primary Care Research Institute in Tarragona, following a simple numerical randomisation ratio. No masking will be possible either for pregnant women or for ASSIR professionals; the data will be masked for the research team carrying out the statistical analyses.

Selection of the participating centres: the pregnancy monitoring centres participating in the recruitment of the study will be four, all of them from the ICS. Three in the Tarragona region (Tarragona, Reus and Valls) and a fourth in the Osona region of Barcelona (Manresa).

Intervention: ASSIR centre will offer treatment, following the standard practice protocols, to all participants who want to quit smoking, following standard practice protocols. Additionally, only participants assigned to the intervention group will have the access code to the Tobbstop App (www.tobbsotop.com) and its use will be recommended. The quality of the intervention will be assured by a three-level control system:

1. Adaptation of the App. The Tobbstop App has been successfully tested in the general population. For the present study the contents will be updated and adapted to the study population (pregnant women). In that sense, a qualitative study will be carried out with the aim of identifying the facilities and barriers that pregnant women face to stop smoking through individual interviews and focus groups.
2. Technical training. Training will be carried out in each of the centres participating in the pregnancy control follow-up visits. The training will be performed by health professionals in order to understand the use of the App.
3. Centralised monitoring. Confirmatory tests will be referred to a single reference observer who will centralise quality control and interpret the results (urinary cotinine).

Follow-up: no additional follow-up visits will be planned for the study. In the scheduled pregnancy follow-up visits, smoking habits will be assessed by a questionnaire and CO level quantification by coximetry. At the end of the pregnancy check-ups, follow-up will be carried out by telephone contact. Women who quit smoking will be scheduled to visit their health centre 12 months after the intervention to find out about their relationship with smoking. If they report abstinence, a coximetry test will be performed and if it is less than 10 ppm (&), urinary cotinine will be determined.

(&) The cut-off point is considered to be 10 ppm, as lower values indicate non-smoking and higher values indicate smoking in the previous 12-24 hours.

Data recording: the information from the study will be recorded in a structured way by a data collection questionnaire and will be stored in an application accessible from the corporate Intranet of the Catalan Institute of Health. Access to this website is restricted and will be controlled by a personal password for each researcher, who will be responsible for entering the records of the participants recruited.

Definition of the outcome variable: prolonged abstinence from drug use will be considered as the main variable, and punctual abstinence as a secondary variable, both validated by biochemical confirmation 12 months after the intervention. Urine cotinine values less than 100ng/ml will reflect an abstinence condition, values between 100 and 500 ng/ml will be accepted as occasional smoker, and values above 500ng/ml will be considered as smoker.

The criteria for establishing abstinence according to the recommendations of the Society for Research on Nicotine and Tobacco:

* Continuous abstinence: sustained abstinence from the time of intervention to a follow-up period.
* Prolonged abstinence: sustained abstinence between an initial grace period ($) and a follow-up period.
* Punctual abstinence: abstinence during a window of time (usually 7 days) immediately preceding the time of follow-up.

($) Grace period is the period immediately following the defined quit date or intervention date in which continued smoking is not counted as failure. For most studies it is recommended to be no longer than 2-4 weeks.

In general, continuous abstinence is accepted as the gold standard. However, this measure is too stringent and prolonged abstinence is preferred as it includes the participants who achierve sustained abstinence after a transitional grace period, which would otherwise be considered failures.

Sample calculation: accepting an alpha risk of 0.05 and a beta risk of less than 0.2 in a bilateral contrast, it will be necessary to include 200 participants in each group, in order to detect the difference between the two proportions statistically significant. In the control group is expected to be 0.5 and in the intervention group 0.65. A loss-to-follow-up rate of 5% is estimated. The ARCSINUS approximation (GRANMO Sample Size Calculator v.7.12 available at www.imim.es) was used.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women smokers (report having smoked sporadically or daily in the last 30 days(*)) over 18 years of age,
* Follow-up of pregnancy in the ASSIR in Camp de Tarragona and Barcelona of the ICS,
* Having a mobile device with Android or iOS operating system and data connection,
* Having skills on the use of Apps and willingness to use them (#).

(*) Active smoking is defined as daily or occasional smoking in the last month, regardless of the amount smoked.

(#) It is understood that you have skills on the use of Apps and willingness to use them if you answer affirmatively to the following questions: Have you downloaded any application on your mobile?, Would you install an application to help you quit smoking on your mobile?, Have you participated in any chat group?, and Have you played any game with your mobile device? (criteria to ensure the usability of the intervention tool).

Exclusion Criteria:

* Having participated in a smoking cessation study within the last 12 months,
* Psychiatric history that prevents or limits follow-up of the study,
* Inability to follow up for any reason,
* Express refusal of the patient to continue in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 400 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Smoking cessation | 1 year
  Women who have stopped smoking during pregnancy will be scheduled to visit their health centre 12 months after the intervention to find out about their relationship with smoking.

SECONDARY OUTCOMES:
Verification of smoking abstinence | 1 year
  If they report abstinence, a coximetry test will be performed and if it is less than 10 ppm (&), a urine sample will be to determine urinary cotinine as a biochemical cessation confirmation.
  (&) The cut-off point is considered to be 10 ppm, as lower values indicate non-smoking and higher values indicate smoking in the previous 12-24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Rey-Reñones, PhD, Principal Investigator — Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Locations (1):
- IDIAP Jordi Gol, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
not yet decided as future studies are being considered and may be considered
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 3 years
Access Criteria: The data will be entered on the IDIAp J Gol institution platform
URL: https://www.idiapjgol.org/index.php/ca/

REFERENCES:
- [Derived] Agras-Guardia M, Martinez-Torres S, Satue E, Granado-Font E, Palleja-Millan M, Patricio D, Leiva M, Rey-Renones C, Martin-Lujan F. Experiences of smoking and tobacco use during pregnancy: A qualitative study protocol. PLoS One. 2024 Aug 9;19(8):e0308781. doi: 10.1371/journal.pone.0308781. eCollection 2024. PMID 39121101
- [Derived] Agras-Guardia M, Martinez-Torres S, Granado-Font E, Palleja-Millan M, Villalobos F, Patricio D, Ruiz F, Marin-Gomez FX, Duch J, Rey-Renones C, Martin-Lujan F. Effectiveness of an App for tobacco cessation in pregnant smokers (TOBBGEST): study protocol. BMC Pregnancy Childbirth. 2022 Dec 13;22(1):933. doi: 10.1186/s12884-022-05250-5. PMID 36514020